CLINICAL TRIAL: NCT03980769
Title: Allogeneic Hematopoietic Cell Transplantation for Patients With Non-Malignant Disorders Using Treosulfan, Fludarabine, and Thiotepa
Brief Title: Donor Stem Cell Transplant With Treosulfan, Fludarabine, and Thiotepa in Treating Patients With Non-malignant Disorders
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1005072; NCI-2019-03243 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9621 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Non-Neoplastic Hematopoietic and Lymphoid Cell Disorder
MeSH Terms: interventions — Thiotepa; treosulfan; fludarabine phosphate; Antilymphocyte Serum; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, transplant) (Experimental): Patients receive thiotepa IV BID over 2 hours on day -7, treosulfan IV over 120 minutes on days -6 to -4, fludarabine phosphate IV over 60 minutes on days -6 to -2, and rabbit anti-thymocyte globulin IV over 4-6 hours on days -4 to -2. Patients then undergo allogeneic hematopoietic cell transplant via infusion on day 0. Patients may also undergo bone marrow biopsy and aspiration and MRI as clinically indicated and blood sample collection on study.
  Interventions: Drug: Thiotepa; Drug: Treosulfan; Drug: Fludarabine Phosphate; Biological: Rabbit Anti-Thymocyte Globulin; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Bone Marrow Biopsy; Procedure: Bone Marrow Aspiration; Procedure: Magnetic Resonance Imaging; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Thiotepa — Given IV
  Other Names: 1,1',1"-phosphinothioylidynetrisaziridine; N,N', N''-Triethylenethiophosphoramid; Oncotiotepa; STEPA; Tepadina; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoramide; Thiotef; Tifosyl; TIO TEF; Triethylene thiophosphoramide; Triethylenethiophosphoramide; TSPA
Drug: Treosulfan — Given IV
  Other Names: (S-(R*,R*))-1,2,3,4-butanetetrol; 1,4-dimethanesulfonate; [R-(R*,S*)]-, 299-75-2, 39069; Dihydroxybusulfan; Ovastat; Treosulphan; Tresulfon
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 312887; 328002; 75607-67-9; 9H-Purin-6-amine; 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; Fludarabine-5'-Monophosphate
Biological: Rabbit Anti-Thymocyte Globulin — Given IV
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo HCT via infusion
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI; MRI Scan
Procedure: Biospecimen Collection — Undergo blood sample collection

SUMMARY:
This phase II clinical trial studies how well treosulfan, thiotepa, fludarabine, and rabbit anti-thymocyte globulin (rATG) before donor stem cell transplantation works in treating patients with nonmalignant (non-cancerous) diseases. Hematopoietic cell transplantation has been shown to be curative for many patients with nonmalignant (non-cancerous) diseases such as primary immunodeficiency disorders, immune dysregulatory disorders, hemophagocytic lymphohistiocytosis, bone marrow failure syndromes, and hemoglobinopathies. Powerful chemotherapy drugs are often used to condition the patient before infusion of the new healthy donor cells. The purpose of the conditioning therapy is to destroy the patient's abnormal bone marrow which doesn't work properly in order to make way for the new healthy donor cells which functions normally. Although effective in curing the patient's disease, many hematopoietic cell transplantation regimens use intensive chemotherapy which can be quite toxic, have significant side effects, and can potentially be life-threatening. Investigators are investigating whether a new conditioning regimen that uses less intensive drugs (treosulfan, thiotepa, and fludarabine phosphate) results in new blood-forming cells (engraftment) of the new donor cells without increased toxicities in patients with nonmalignant (non-cancerous) diseases.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive thiotepa intravenously (IV) twice daily (BID) over 2 hours on day -7, treosulfan IV over 120 minutes on days -6 to -4, fludarabine phosphate IV over 60 minutes on days -6 to -2, and rabbit anti-thymocyte globulin IV over 4-6 hours on days -4 to -2. Patients then undergo allogeneic hematopoietic cell transplant via infusion on day 0. Patients may also undergo bone marrow biopsy and aspiration and magnetic resonance imaging (MRI) as clinically indicated and blood sample collection on study.

After completion of study treatment, patients are followed up at 1 year and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patient with nonmalignant disease treatable by allogeneic HCT
* Patient with a nonmalignant disease that is not clearly defined (a patient with a non-malignant disease for whom genetic testing has been done and a genetic mutation responsible for their non-malignant disease phenotype has not been identified) are eligible for the study following discussion with and approval by the protocol principal investigator (PI) (Dr. Lauri Burroughs)
* Age < 50 years
* DONOR: Human leukocyte antigen (HLA)-identical related donor OR unrelated donor matched for HLA-A, B, C, DRB1 and DQB1 or mismatched for a single allele at HLA-A, B, C, or a single DQB1 antigen or allele mismatch by high resolution deoxyribonucleic acid (DNA) typing
* DONOR: Bone marrow is the preferred cell source (when feasible). However, peripheral blood stem cells (PBSC) is also allowed and the PI may determine if PBSC is preferred for certain patients

  * The recommended total nucleated cell count (TNC) for bone marrow grafts is >= 4.0 x 10^8 TNC/kg (actual recipient weight)
  * The recommended CD34 cell count for PBSC grafts is >= 5 x 10^6 CD34/kg (actual recipient weight) and the recommended maximum CD34 cell count for PBSC grafts is 10 x 10^6 CD34/kg (actual recipient weight)
* DONOR: HLA-matched sibling bone marrow in combination with HLA-matched sibling umbilical cord blood if the HLA-matched sibling umbilical cord blood was collected and stored. The HLA-matched sibling bone marrow and cord blood would be matched for HLA-A, B, C, DRB1 and DQB1

Exclusion Criteria:

* Patients with idiopathic aplastic anemia and Fanconi anemia; patients with aplastic anemia associated with paroxysmal nocturnal hemoglobinuria (PNH) or inherited marrow failure syndromes (except Fanconi anemia) will be allowed
* Impaired cardiac function as evidenced by ejection fraction < 35% (or, if unable to obtain ejection fraction, shortening fraction of < 26%) or cardiac insufficiency requiring treatment or symptomatic coronary artery disease. Patients with a shortening fraction of < 26% may be enrolled if approved by a cardiologist
* Impaired pulmonary function as evidenced by carbon monoxide diffusing capability (DLCO) corrected < 50% of predicted (or, if unable to perform pulmonary function tests, then oxygen [O2] saturation < 92% on room air)
* Impaired renal function as evidenced by:

  * Estimated creatinine clearance < 60 mL/min/1.73m^2 using either the Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) equation for adult patients (>= 18 years old), or the updated Schwartz formula for pediatric patients (< 18 years old). If the estimated creatinine clearance is < 60 mL/min/1.73m^2, then renal function must be measured by 24-hour creatinine clearance, Iothalamate, Iohexol or nuclear GFR and the patient is excluded if their measured creatinine clearance is < 50 mL/min/1.73 m^2, OR
  * Serum creatinine > 2 x upper limit of normal, OR
  * Dialysis dependent
* Evidence of synthetic dysfunction or severe cirrhosis requiring deferral of conditioning as recommended by a gastroenterology specialist
* Active infectious disease requiring deferral of conditioning as recommended by an infectious disease specialist
* Positive for HIV (human immunodeficiency virus)
* Females who are pregnant or breast-feeding
* Known hypersensitivity to treosulfan, fludarabine, and/or thiotepa
* DONOR: Donors deemed unable to undergo marrow harvesting of PBSC mobilization and leukapheresis
* DONOR: HIV-positive donors
* DONOR: Donors with active infectious hepatitis
* DONOR: Female donor with positive pregnancy test
* DONOR: Donors are excluded if the patient has an identified antibody against a donor-specific HLA locus as specified in standard practice
* DONOR: HLA-matched sibling cord blood units that have not passed donor screening for infectious disease markers as recommended by the National Marrow Donor Project (NMDP) will not be used unless a waiver is signed by the clinical attending allowing use of cord blood unit. Cord blood units are presumed to be cytomegalovirus (CMV) negative regardless of serologic testing due to passive transmission of maternal CMV antibodies

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Engraftment failure | 1 year after transplant
  Will be defined as donor CD3 chimerism < 5% at 1 year after transplant.

SECONDARY OUTCOMES:
Overall survival | At 1 year post-transplant
Event-free survival | At 1 year post-transplant
  Defined as death due to any cause, donor lymphocyte infusion, CD34 boost, second transplant, graft rejection or graft failure, or the development of myelodysplastic syndrome or leukemia following transplant (whichever event occurs first).
Transplant-related mortality | At day 100 after transplant
Incidence of grade II-IV acute graft-versus-host disease | At day 100 after transplant
Incidence of chronic graft-versus-host disease | At 1 year after transplant
Donor chimerism CD3 & CD33 | At 1 year after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Lauri Burroughs, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No